CLINICAL TRIAL: NCT04512586
Title: Physiological Pacemaker Treatment in Combination With AV Node Ablation Compared With Pulmonary Vein Isolation for Patients With Symptomatic Atrial Fibrillation - a Randomized Controlled Study
Brief Title: His-pacing and AV-node Ablation vs. Pulmonary Vein Isolation for Atrial Fibrillation
Acronym: His-PAAF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment too slow. Unrealistic to finish study with full inclusion cohort.
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: His_PAAF_study
Record Dates: First submitted 2020-07-01; First posted 2020-08-13 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Left Atrial Dilatation
Keywords: Atrial fibrillation; Left atrial dilatation; Pulmonary vein isolation; AV node ablation; Conduction System pacing; Quality of Life; Age group 70 to 85 years
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients are randomized to either
  1. Conduction system pacing via His-pacing electrode, in combination with AV node ablation
  2. Pulmonary vein isolation ablation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conduction System pacing plus AV node ablation (Experimental): A His-pacing lead in combination with a backup RV pacing lead or an LBB pacing lead, and a right atrial lead (if needed) will be placed using standard technique. The His-pacing or LBB pacing lead will be Medtronic 3830, and the outer sheath will be either Medtronic C304 or C315 deflectable. If failure to implant with these tools, other leads and sheaths can be used at the discretion of the operator. A standard DDD pacemaker or CRT-P device from Medtronic will be used.
  A minimum of three weeks post-implant, the device will be interrogated and His-bundle threshold will be evaluated. A threshold of ≤2.0V@1.0ms is acceptable. If the device is well-functioning and successful His-pacing is documented, AV node ablation will be performed.
  Interventions: Procedure: Conduction System pacing and AV node ablation
- Pulmonary vein isolation (Active Comparator): Atrial fibrillation will be performed as a complete pulmonary vein isolation. Either Cryoballon or radio frequency ablation with irrigated tip contact force enabled catheter can be used. Pulsed field ablation can be used if available. Endpoint is complete electrical isolation of all pulmonary veins, verified by entry- and exit block using a multipolar catheter during pacing.
  Interventions: Procedure: Atrial fibrillation ablation by pulmonary vein isolation

INTERVENTIONS:
Procedure: Conduction System pacing and AV node ablation — See study arm description.
  Arms: Conduction System pacing plus AV node ablation
Procedure: Atrial fibrillation ablation by pulmonary vein isolation — See study arm description
  Arms: Pulmonary vein isolation

SUMMARY:
Objective To investigate if conduction system pacing ((CSP) i.e. atrioventricular node ablation + His bundle pacing or Left Bundle Branch pacing) is as good as (or better than) atrial fibrillation ablation with pulmonary vein isolation for older patients (70-85yrs) with symptomatic atrial fibrillation and at least moderately dilated left atrium.

Patient population:

90 patients aged 70-85 years with atrial fibrillation, referred to either AV node ablation or pulmonary vein isolation.

Primary endpoint:

Improvement in health-related quality of life as measured by the physical component summary (PCS) of the well-validated SF-36 form, at one year after AV node ablation + CSP or AF ablation.

Secondary endpoints:

Physical performance measured by 6-minute walk test, biochemical markers of heart failure (NT-ProBNP), frequency of complications, left ventricular systolic and diastolic function, and left atrial size evaluated after 12 months. Arrhythmia specific symptoms and anxiety will be measured with the ASTA and HADS questionnaires. Arrhythmia symptom correlation between subjective and objective findings. After three years, clinical endpoints will be evaluated regarding overall survival, and risk of heart failure hospitalization or death. The cost of the treatments will be compared, and estimated cost per quality adjusted year of life will be calculated, based on the EQ5D questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Indication for invasive treatment of symptomatic atrial fibrillation according to current guidelines
* LVEF >35%
* Age 70-85 years
* Persistent atrial fibrillation, or paroxysmal atrial fibrillation with at least moderate enlargement of the left atrium (≥42ml/m2)
* Chronic and well-tolerated treatment with anticoagulants (either non-vitamin K oral anticoagulant or vitamin K antagonist)
* Willingness to participate, to understand the instructions and fill out the questionnaires, and ability to sign informed consent

Exclusion Criteria:

* Chronic atrial fibrillation with >1 year duration
* BMI >40kg/m2
* Hypertrophic cardiomyopathy
* Severe heart failure with symptoms ≥ NYHA class IIIb
* Heart amyloidosis
* Cardiac sarcoidosis
* Recent (<3 months) myocardial infarction
* Significant heart valve disease (pronounced insufficiency or stenosis)
* Pacemaker or ICD treatment ongoing, or current pacemaker indication
* Congenital heart disease that required surgical correction
* Comorbidity that is assessed significantly affect the patient's quality of life over the next year, or 3-year survival

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Health related Quality of Life: questionnaire | 12 months
  Improvement in the Physical Component Summary (PCS) of the SF-36 questionnaire

SECONDARY OUTCOMES:
Safety endpoint: Proportion of patients with major adverse events | 12 months
  Proportion of patients with major adverse events that are devicerelated or related to ablation procedure (including but not limited to exit block, infection, perforation/tamponade, pericardial effusion, lead dislodgement, TIA/stroke, oesophago-atrial fistula, groin hematoma or vascular complication, pseudoaneurysm, phrenic nerve injury).
Mental Quality of Life: questionnaire | 12 months
  Improvement of the "mental" health related quality of life, measured by the mental component summary (MCS) of the SF-36 questionnaire
Arrhythmia related Quality of Life: ASTA questionnaire | 12 months
  Change in arrhythmia related quality of life as measured by the The Arrhythmia-Specific questionnaire in Tachycardia. The ASTA questionnaire consists of 13 items, each with a score of 0-4. A higher score denotes more symptoms associated with the arrhythmia.
  and Arrhythmia (ASTA) questionnaire
Anxiety and depression | 12 months
  Anxiety and depression symptoms, measured by the Hospital Anxiety and Depression Scale (HADS). The scale consists of 14 questions with 0 to 3 points for each, with a higher score denoting more depression/anxiety
Ejection fraction | 12 months
  Change in left ventricular systolic ejection fraction
Biomarker for heart failure | 12 months
  Change in NT-ProBNP level
Physical performance | 12 months
  Change in six minute walk test distance
Electrocardiography changes | 12 months
  Change in QRS duration on ECG
Health economy | 12 months
  Total atrial fibrillation and device related health care cost
Survival | 3 years
  Total survival and survival free of major complications
Hospitalization for heart failure | 3 years
  Risk of hospitalization for heart failure assessed by Kaplan Meier time dependent analysis using time from ablation to first hospitalization for heart failure within three years

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Borgquist, MD PhD, Principal Investigator — Lund University, Skane University Hospital, Arrhythmia Section, Lund, Sweden
Locations (4):
- Sweden (4):
  - Linköping University, Linköping
  - Skane University Hospital, Lund
  - Stockholm Arrhythmia Center, Stockholm
  - Varberg Hospital, Varberg

IPD SHARING:
Plan to Share IPD: No